CLINICAL TRIAL: NCT03487081
Title: Neural Predictors of Social Emotion Regulation Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Kevin Ochsner, Professor of Psychology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: AAAR8654; R01AG043463 (NIH)
Record Dates: First submitted 2018-03-22; First posted 2018-04-03 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Emotions; Rumination
MeSH Terms: conditions — Rumination Syndrome | interventions — Social Control, Formal; Professional Autonomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social regulation (Experimental): Following the fMRI session, participants in the social regulation group will be asked to rate their mood twice a day for 3 weeks. Furthermore, every other day, they will receive one event written by another participant. They will be asked to help the other person use emotion regulation strategies to feel less negative. The participant will answer brief questions related to his/her feelings after receiving the event and after providing social emotion regulation.
  Interventions: Behavioral: Social regulation
- Self regulation (Active Comparator): Following the fMRI session, participants in the self regulation group will be asked to rate their mood twice a day for 3 weeks. Furthermore, every other day, they will write an event that caused them negative emotions. They will be asked to use emotion regulation strategies to decrease their negative emotions. The participant will answer brief questions related to his/her feelings after writing the event and after implementing the emotion regulation strategy.
  Interventions: Behavioral: Self regulation

INTERVENTIONS:
Behavioral: Social regulation — Participants will be instructed to help another person think about their negative events differently using an emotion regulation strategy called reappraisal.
  Arms: Social regulation
Behavioral: Self regulation — Participants will be instructed to think about their negative events by reframing the meaning of the event. This is a typical strategy in emotion regulation research known as reappraisal.
  Arms: Self regulation

SUMMARY:
The purpose of this study is to investigate the basic psychological and neural mechanisms underlying the social regulation of emotion - that is, how one person's actions can impact, or regulate - the emotions of another person - and how this ability changes with practice. As such, this study is not designed to directly address clinical health outcomes and provide no treatment or intervention.

DETAILED DESCRIPTION:
Prior research has demonstrated that helping others regulate their emotions has benefits for the support provider. But little is known about the basic brain mechanisms underlying this ability or how this ability can change with practice. To address these questions, this study has two parts. In the first, functional magnetic resonance imaging (fMRI) is used to gain insight into the brain systems involved in helping others regulate negative emotions by comparing them to the brain systems involved in regulating the participants' own negative emotions. In the second part, participants engage in three weeks of structured practice, or training, in either socially regulating others' emotions or in self-regulating their own emotions. The investigators predict that helping others regulate their emotions will involve many of the same brain regions implicated in regulating one's own emotions, in addition to regions involved in perspective taking and the reward of helping others. Further, when relating the brain data from part 1 to the regulation practice data from part 2, the investigators expect that individuals who in part 1 show greater activity in brain regions supporting either social or self-regulation may be more likely in part 2 to show corresponding improvements in regulation performance. The results of these studies are intended to lay the groundwork for future studies investigating the social regulation of emotion in older adults and clinical populations for whom social support can be beneficial.

ELIGIBILITY:
Inclusion Criteria:

* Native English speaker
* Right handed

Exclusion Criteria:

* Current or past history of neurological or psychiatric illness
* Use of psychoactive drugs
* Individuals who have metal devices or implants that cannot be removed from their body (e.g., piercings, pacemakers, copper intrauterine devices (IUDs))
* Pregnant women

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2019-02-11 (Actual); Study Completion 2019-02-11 (Actual)

PRIMARY OUTCOMES:
Emotion Regulation Questionnaire (ERQ) Score | Change from baseline at 3 weeks follow up
  The Emotion Regulation Questionnaire (10 items) has 2 subscales - suppression and reappraisal. Participants rate their response on a 7-point Likert scale ranging from 1 (Strongly disagree) to 7 (Strongly agree). The total score is calculated from the sum of the items in each subscale. Higher scores indicate higher tendency to use the emotion regulation strategy.
Ruminative Response Scale (RRS) Score | Change from baseline at 3 weeks follow up
  The Ruminative Response Scale (22 items) has 3 subscales - brooding, reflection and depression. Participants rate their response on a 4-point Likert scale ranging from 1 (Almost never) to 4 (Almost always). The total score is calculated from the sum of the items in each subscale. Higher scores indicate higher tendency to engage in ruminative thoughts.

SECONDARY OUTCOMES:
Change in mood rating (Likert scale score) | Baseline, up to 3 weeks
  Participants rate their response indicating their current emotions (e.g., angry, happy, sad) on a 9-point Likert scale ranging from 1 (completely disagree) to 9 (completely agree). The total score for positive mood is calculated from the sum of 4 positive emotion items. The total score for negative mood is calculated from the sum of 4 negative emotion items.
Change in Brief State Rumination Inventory (BSRI) (Likert scale score) | Baseline, up to 3 weeks
  Participants rate their response indicating their ruminative thought (e.g., "Right now, I wonder why I react the way I do") on a 9-point Likert scale ranging from 1 (completely disagree) to 9 (completely agree). The total score is calculated from the sum of all 13 items.
State Trait Anxiety Inventory (STAI) - Trait Scale (Likert scale score) | Change from baseline at 3 weeks follow up
  The State Trait Anxiety Inventory - Trait scale (20 items) measures trait anxiety. Participants rate their response on a 4-point Likert scale ranging from 1 (Almost never) to 4 (Almost always). The total score is calculated from the sum of all items. Higher scores indicate higher anxiety.
Center for Epidemiologic Studies Depression Scale (CES-D) (Likert scale score) | Change from baseline at 3 weeks follow up
  The Center for Epidemiologic Studies Depression Scale (20 items) measures depression. Participants rate their response on a 4-point Likert scale ranging from 0 (Rarely or none of the time (less than 1 day)) to 3 (All of the time (5-7 days)). The total score is calculated from the sum of all items. Higher scores indicate higher depression level.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Ochsner, PhD, Principal Investigator — Department of Psychology, Columbia University
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided